CLINICAL TRIAL: NCT06702969
Title: Influence of Digitalized Impression on Single Peri-implant Soft Tissue Profile in Esthetic Zone and Patient Satisfaction: A Randomized Controlled Trial
Brief Title: Influence of Digitalized Impression on Single Peri-implant Soft Tissue Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Digitalized Impression
Record Dates: First submitted 2024-11-03; First posted 2024-11-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2023-01

CONDITIONS: Patient Satisfaction
Keywords: Immediate implant; Digital impression; Pink esthetic score; Conventional impression
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital impression with intraoral scanner (Active Comparator): included seven participants with non-restorable tooth in esthetic zone replaced by immediate implants receiving a single all ceramic crown fabricated with full digital procedure consisting of digital impression with intraoral scanner, and Computer Aided Design/ Computer Aided Manufacture (CAD/CAM) procedure.
  Interventions: Device: Intra oral scanner
- conventional impression technique (Active Comparator): included seven participants with non-restorable tooth in esthetic zone replaced by immediate implants receiving a single all ceramic crown fabricated with Conventional impression-taking with polyvinyl siloxane, plaster model pouring and lost-wax casting technique
  Interventions: Device: impression analog

INTERVENTIONS:
Device: Intra oral scanner — Immediate implant placement with customized healing abutment and after three months placement all ceramic crown by digital impression using intra oral scanner
  Other Names: implant placement
  Arms: Digital impression with intraoral scanner
Device: impression analog — Immediate implant placement with customized healing abutment and after three months placement of all ceramic crowns by conventional impression
  Other Names: implant placement; impression copying
  Arms: conventional impression technique

SUMMARY:
This randomized controlled clinical study will be carried out to compare the digital with conventional impression procedures for the restoration of single implants in an esthetic zone by assessing:

1. pink esthetic score (PES) of peri-implant soft tissue profile and marginal bone loss (MBL) as primary objectives
2. Patients' satisfaction and clinical outcomes as secondary objectives

DETAILED DESCRIPTION:
fourteen patients with single nonrestorable tooth in the esthetic zone participated in the study and were replaced with immediate implants with immediate customized provisional restoration after 3 months they recalled for the impression, seven with digital and the others with conventional and evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders within age range of 20-50 years.
2. Systemically healthy participants classified as American Society of Anesthesiologists( ASA ) class I . Guided by medical questionnaire modified from Burkett's
3. Single non restorable tooth in upper anterior esthetic zone with at least 4 mm bone present apical to the root apex for primary stability.
4. Type I extraction sockets according to classification.
5. Ability to attend the surgery , comply to it's procedures , the recall visits and oral hygiene protocol .
6. Thick gingival phenotype with thickness ≥ 2 mm around the non-restorable tooth -

Exclusion Criteria:

1. Missing adjacent teeth or opposing tooth. .
2. Acute periapical pathosis or active periodontal infections related to non-restorable tooth or adjacent teeth.
3. Smokers.
4. Pregnant or lactating females.
5. Patients with para-functional habits (bruxism and/or clenching)
6. Vulnerable groups (handicapped, orphans, and prisoners). -

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
pink esthetic score | at the baseline(time of impression), second time was one week later (immediately) after crown placement, third time was one month later after crown placement , fourth time was three months later after crown placement
  The pink esthetic score is based on seven variables:
  * Mesial papilla
  * Distal papilla
  * Soft-tissue level
  * Soft- tissue contour
  * Alveolar process deficiency
  * Soft-tissue color and texture Each variable was assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score
marginal bone loss | immediately after crown placement (baseline), then three months after crown placement
  described by millimeter using paralleling technique

SECONDARY OUTCOMES:
patient satisfaction | after crown placement
  satisfaction questionnaire modified from based on 10 specific questions.
  The questions were as follows:
  1. Are you satisfied with the treatment? with 0 = very dissatisfied and 100 = very satisfied
  2. Did you experience discomfort during the impression-taking? with 0 = high discomfort and 100 = no discomfort
  3. Did you experience gag reflex/nausea during the impression-taking? with 0 = strong gag reflex/nausea, and 100 = no gag reflex/nausea
  4. How comfortable was the impression procedure? with 0 = uncomfortable and 100 = comfortable
  5. Does your implant-supported restoration function well? with 0 = bad function and 100 = well function
plaque index | Immediately after crown placement (baseline), one months later , and finally three months after crown placement
  0 = No plaque in gingival area.
  1. = A film of plaque adhering to the free gingival margin and adjacent area of tooth. The plaque may be recognized only by running a probe across the tooth surface.
  2. = Moderate accumulation of soft deposit within the gingival pocket and on the gingival pocket and on the gingival margin and/or adjacent tooth surface that can be seen by naked eye.
  3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
     * of sites positive for dental plaque will be calculated for each case.
gingival index | Immediately after crown placement (baseline), one months later , and finally three months after crown placement
  0 = Normal gingiva.
  1. = Mild inflammation, slight change in color, slight edema; no bleeding on probing.
  2. = Moderate inflammation, redness, edema, and glazing; bleeding on probing.
  3. = Sever inflammation, marked redness and edema, ulceration; tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: ola A ezzat, professsor, Study Director — faculty of dentistry-Ain shams university
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No